CLINICAL TRIAL: NCT06462846
Title: Evaluation of Demographic and Clinical Characteristics and Intraoperative and Pathological Findings in Patients With Suspected Appendicitis Who Underwent Appendectomy in 5 Azar Hospital in 2022
Brief Title: Evaluation of Clinical Characteristics and Pathological Findings in Patients With Suspected Appendicitis
Status: Completed | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, ronak jalali, Medical student, Golestan University of Medical sciences
Other Study IDs: 113867
Record Dates: First submitted 2024-06-01; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Appendicitis
Keywords: Appendicitis; Appendectomy; Appendicitis diagnosis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As we know, one of the most common reasons for people to visit health centers and hospitals (15%) is abdominal pain, and appendicitis is at the top of their diagnosis in the 2-4th decade of age, which in most cases For treatment, considering the patient's condition and the need for surgery, appendectomy is the first method. One of the things that helps us a lot in this area is the epidemiology and incidence of this disease in the target society, which sometimes varies in different regions. One of the things that can be checked in this disease is the age and gender of the person and its incidence in different age ranges.

DETAILED DESCRIPTION:
appendicitis is one of the most important reasons for people to go to the hospital, and 15% of the visits to the hospital are for this reason, and sometimes patients end up undergoing appendectomy. The mortality rate of this disease is 0.2-1% among young people and 8% among people over 65 years old In some people, depending on the sex, age, pregnancy and related diseases and even the weight of the people, the location of the appendix is different and this issue is very important during surgery. Different positions of the appendix, such as retro-scapular, subhepatic, pelvic, etc., create different challenges during surgery, so investigating the possibilities of the location of the appendix is an important issue in the decision-making and preparation of the patient and the surgical team.

Also, laboratory criteria such as wbc, diff, plt, crp can also help in diagnosing this disease. In this project, in addition to the above, the chief complaints and accompanying symptoms of people have also been examined

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of appendicitis
* appendectomy

Exclusion Criteria:

* Lack of required information in medical documents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patents operated with the diagnosis of appendicitis in 5th azar medical center, in 2022
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The accuracy of imaging in determining the size of the appendix in patients with suspected appendicitis | One year
  comparison of the appendix size reported in radiologic studies with pathologic findings

SECONDARY OUTCOMES:
correlation between CRP levels and pathologic findings in patients with suspected appendicitis | One year
  Comparison of CRP levels in the different stages of appendicitis according to pathologic reports
correlation between WBC measures and pathologic findings in patients with suspected appendicitis | One year
  Comparison of WBC measures in the different stages of appendicitis according to pathologic reports
sex distribution in patients with suspected appendicitis | one year
  the prevalence and percentage of each sex group in patients with suspected appendicitis
Age distribution in patients with suspected appendicitis | one year
  the prevalence and percentage of each age group in patients with suspected appendicitis
prevalence of clinical findings in patients with suspected appendicitis | one year
  prevalence and percentage of each clinical finding (fever, anorexia, shifting pain, tenderness, rebound tenderness, rovsing sign, psoas sign) in patients with suspected appendicitis

CONTACTS AND LOCATIONS:
Locations (1):
- Golestan University of Medical Sciences, faculty of medicine, Gorgan, Golestan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JH, Park YS, Choi JS. The epidemiology of appendicitis and appendectomy in South Korea: national registry data. J Epidemiol. 2010;20(2):97-105. doi: 10.2188/jea.je20090011. Epub 2009 Dec 19. PMID 20023368
- [Background] Golz RA, Flum DR, Sanchez SE, Liu X, Donovan C, Drake FT. Geographic Association Between Incidence of Acute Appendicitis and Socioeconomic Status. JAMA Surg. 2020 Apr 1;155(4):330-338. doi: 10.1001/jamasurg.2019.6030. PMID 32129808
- [Background] Tavra A, Quien D, Barcot O. Oncological aspect of incidental appendectomy with regard to histopathological findings: A retrospective cohort study. Eur J Surg Oncol. 2023 Oct;49(10):107013. doi: 10.1016/j.ejso.2023.107013. Epub 2023 Aug 11. PMID 37597285
- [Background] Yagmur Y, Sogutcu N, Gumus S. Recent classifications systems for gastroenteropancreatic neuroendocrine tumors A single-center experience. Ann Ital Chir. 2020;91:598-604. PMID 32989209
- [Background] Bayhan Z, Yildiz YA, Akdeniz Y, Gonullu E, Altintoprak F, Mantoglu B, Capoglu R, Kahyaoglu Akkaya Z. Appendix Neuroendocrine Tumor: Retrospective Analysis of 4026 Appendectomy Patients in a Single Center. Emerg Med Int. 2020 Sep 3;2020:4030527. doi: 10.1155/2020/4030527. eCollection 2020. PMID 32963833
- [Background] Henriksen SR, Rosenberg J, Fonnes S. Other Pathologies Were Rarely Reported after Laparoscopic Surgery for Suspected Appendicitis: A Systematic Review and Meta-Analysis. Dig Surg. 2023;40(3-4):91-99. doi: 10.1159/000531283. Epub 2023 Jul 18. PMID 37463567
- [Background] Jukic M, Nizeteo P, Matas J, Pogorelic Z. Trends and Predictors of Pediatric Negative Appendectomy Rates: A Single-Centre Retrospective Study. Children (Basel). 2023 May 15;10(5):887. doi: 10.3390/children10050887. PMID 37238435
- [Result] Pineda Villeda RH, Flores Reyes DL, Suazo Rivera JF. Acute Appendicitis: Epidemiological, Clinical, Surgical, and Post-surgical Characteristics in a Honduran General Hospital. Cureus. 2023 Jun 14;15(6):e40428. doi: 10.7759/cureus.40428. eCollection 2023 Jun. PMID 37456484